CLINICAL TRIAL: NCT04548817
Title: Prospective Registry of Patients With Neurocutaneous Melanocytosis (NCM) Including Cutaneous and CNS Involvement
Brief Title: Neurocutaneous Melanocytosis Registry
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-363
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cutaneous Melanocytic Neoplasm; Large Cutaneous Melanocytic Nevi; Neurocutaneous Melanocytosis
Keywords: large cutaneous melanocytic nevi; LCMN; neurocutaneous melanocytosis; NCM; 20-363; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Neurocutaneous melanosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurocutaneous Melanocytosis: Participants will have Neurocutaneous Melanocytosis (NCM) Including Cutaneous and CNS Involvement

SUMMARY:
This study will involve collecting information about the regular medical care you receive for large cutaneous melanocytic nevi (LCMN) or neurocutaneous melanocytosis (NCM).

ELIGIBILITY:
Inclusion Criteria:

* Patients with LCMN, defined as:

  * Dark-colored patch of skin present at birth
  * Can be located anywhere on the individual's skin
  * May include satellite lesions
  * May be associated with hypertrichosis

OR, in absence of cutaneous involvement:

* histologically or radiographically confirmed CNS melanocytosis.

  * Any age at diagnosis.
  * Signed informed consent by a patient, or parent/legal guardian.
  * Deceased patients can be included provided that parent/legal guardian is contacted at least 6 months after the death of the child and not on the child's birthday or anniversary of death.

Pathology review at MSK is not mandatory to confirm the diagnosis of LCMN or NCM. We will not require pathology analysis of leptomeningeal deposits in patients where characteristic skin lesions are present and melanosis of the meninges is radiographically evident. However, if pathology samples have already been obtained as part of a patient's evaluation and treatment at another institution, tissue samples will be requested for review and confirmation of the diagnosis.

Exclusion Criteria:

* Informed consent has not been provided.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A target sample of 75 patients with LCMN and/or NCM will be enrolled in this registry study. The study is expected to accrue over ≥ 7 years. Currently, an estimated 50 LCMN patients are followed at MSK and we anticipate 25 or more to be referred from outside providers or from new patients seen at MSK. The patient population and the MSK referral base is growing at this time, making this enrollment goal as feasible.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2027-09-03 (Estimated); Study Completion 2027-09-03 (Estimated)

PRIMARY OUTCOMES:
Collect retrospective and prospective clinical, treatment and outcome data about patients with Neurocutaneous Melanocytosis (NCM) worldwide | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Khakoo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Boston Children's Hospital (Data Analysis Only), Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org